CLINICAL TRIAL: NCT00450554
Title: EVALUATION DE LA REPONSE IMMUNITAIRE CONTRE LA SOUCHE DE NEISSERIA MENINGITIDIS B:14,P1.7,16
Brief Title: Immunogenicity After Two Doses of Meningococcal Outer Membrane Vesicle Vaccine MenBVac
Status: Completed | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2007/004/HP
Record Dates: First submitted 2007-03-19; First posted 2007-03-22 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2012-03

CONDITIONS: Vaccination
Keywords: Neisseria meningitidis B:14, P1-7, 16; Serum bactericidal activity; Menbvac

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The main objective of the study is to estimate the proportion of children, born between the 01/01/2002 and the 06/23/200, living around Dieppe (cantons Dieppe est, Dieppe Ouest and Offranville), vaccinated by MenBVac, with a serum bactericidal activity against B:14,P1-7,16 clone related to a protection (>= 4), before and after the third MenBvac vaccination.

ELIGIBILITY:
Inclusion Criteria:

* children born between 01/01/2000 and 06/23/2005, living in Dieppe-Est, Dieppe-Ouest and Offranville, vaccinated twice by MenBVac
* parental authority(ies)assent

Exclusion Criteria:

* no parental authority(ies)assent
* no blood sample during the third vaccination
* impossibility of third vaccination

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: children born between 01/01/2000 and 06/23/2005, living in Dieppe-Est, Dieppe-Ouest and Offranville
Sampling Method: Probability Sample
Enrollment: 236 (Actual)
Dates: Start 2007-02; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: CARON François, Professor, Principal Investigator — Service des Maladies Intectieuses et Tropicales
Locations (1):
- UH-rouen, Rouen, Seine Maritime, France